CLINICAL TRIAL: NCT06320730
Title: Impact of Glycemic Control After Reperfusion on Acute Kidney Injury in Living Donor Liver Transplantation: A Propensity Score-matched Analysis
Brief Title: Impact of Glycemic Control After Reperfusion on Acute Kidney Injury in Living Donor Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jun-Gol Song, Professor, Asan Medical Center
Other Study IDs: 2020-0675
Record Dates: First submitted 2024-03-08; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Acute Kidney Injury; Hyperglycemia; Hypoglycemia; End Stage Liver Disease
MeSH Terms: conditions — Acute Kidney Injury; Hyperglycemia; Hypoglycemia; End Stage Liver Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 110 < REP BG < 180: Those with blood glucose levels over 110 and under 180 after reperfusion in liver transplantation recipients.
  Interventions: Other: Observational study, records of blood glucose level after reperfusion
- Group REP BG ≤110 or ≥180: Those with blood glucose levels below 110 or above 180 after reperfusion in liver transplantation recipients.

INTERVENTIONS:
Other: Observational study, records of blood glucose level after reperfusion — Analyzes blood glucose level after reperfusion by dividing it into two groups: those with blood glucose levels between 110 and 180 and those with blood glucose levels below 110 or above 180.
  Groups: Group 110 < REP BG < 180

SUMMARY:
This retrospective cohort study of patients classified by the blood glucose level after reperfusion in liver transplantation repicient. Our object is to investigate whether controlling BG levels within the optimal range during neohepatic phase is associated with a reduction of AKI incidence. Furthermore, severe AKI, chronic kidney disease (CKD), major adverse cardiac event (MACE) and mortality were also investigated.

DETAILED DESCRIPTION:
The detrimental impact of glucose instability including hyper- and hypoglycemia on postoperative outcomes has been well-established in various fields, particularly in cardiac surgery, and intensive care unit settings. Also, glucose instability occurs frequently in liver transplantation (LT) surgery, attributed to factors such as insulin resistance, surgical stress, and onset of gluconeogenesis after reperfusion of the newly transplanted graft. Previous reports have demonstrated that hyperglycemia is associated with increased mortality, a higher incidence of graft rejection, and surgical site infection in LT. Alongside hyperglycemia, it is also important to consider hypoglycemia, given its association with adverse outcomes.

Acute kidney injury (AKI) stands as one of the most common and critical complications following LT, impacting extended duration of hospital stay, increased morbidity, and mortality. Although the etiology of AKI after LT is multifactorial, perioperative hyper- and hypoglycemia have also been suggested as potential risk factors for postoperative AKI. However, a recent study only has demonstrated that increased glucose variability, rather than hyper-and hypoglycemia alone, is associated with postoperative AKI after LT. The contradictory results observed to date may be attributed to differences in the definition of hyperglycemia, reflecting the challenges in determining the optimal blood glucose (BG) level in LT. In our study, the optimal BG level was determined according to the most recently updated and professional guidelines on glycemic control.

Identifying the timing for glycemic control during LT is also as crucial as determining the optimal BG level. BG levels reach their peak in the neohepatic phase and begin to decrease 3 hours after reperfusion. This excessively elevated hyperglycemia is due to glucose influx from the grafted liver, in addition to peripheral insulin resistance, and gradually decreases after successful LT. Therefore, maintaining a well-controlled BG level within the optimal range, especially during the neohepatic phase, may be associated with better outcomes after transplantation.

Our object is to investigate whether controlling BG levels within the optimal range during neohepatic phase is associated with a reduction of AKI incidence. Furthermore, severe AKI, chronic kidney disease (CKD), major adverse cardiac event (MACE), and mortality were also investigated.

ELIGIBILITY:
Inclusion Criteria:

* Living donor liver transplantation recipients

Exclusion Criteria:

* The exclusion criteria were as follows: recipients under 18 years old, recipients who had undergone deceased donor liver transplantation, recipients who had undergone re-transplantation, recipients with impaired renal function such as CKD or HRS, or those with insufficient data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: living donor liver transplant recipients at Asan Medical Center, Seoul, Korea, Republic of Korea, from January 2008 to December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 3790 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
incidence of acute kidney injury | within 7 days after surgery
  determined by change in sCr according to the Kidney Disease: Improving Global Outcomes (KDIGO) definition (increase in sCr of ≥26.5 mmol litre-1 within 48h or ≥1.5 times baseline within 7 days after surgery)

SECONDARY OUTCOMES:
incidence of severe AKI | within 7 days after surgery
  Severe AKI was defined as KIDIGO stage 2 or 3
incidence of chronic kidney disease (CKD) | within 1 year after surgery
  when renal function assessed by calculating estimated serum glomerular filtration using the abbreviated modification of diet in renal disease equation was <60 mL/min/1.73 m2 for 3 months or more, irrespective of cause
incidence of Major adverse cardiac event (MACE) | within postoperative 30 days (POD30)
  MACE was defined including myocardial infarction (MI), atrial fibrillation (AF), pulmonary thromboembolism (PTE), heart failure (HF), cardiac arrest, and/or stroke
overall mortality | the mortality at overall period (calculated from the date of surgery to the last follow-up) from the date of surgery (up to 10 years)
  overall mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Jun-Gol Song, Seoul, Song-pa Gu, South Korea

IPD SHARING:
Plan to Share IPD: No